CLINICAL TRIAL: NCT04527120
Title: Indigenously Developed Ultrasound Phantom Model vs a Commercially Available Training Model: a Randomised Triple Blind Study
Brief Title: Indigenously Developed Ultrasound Phantom Model
Acronym: IDUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Siju V Abraham, MD, Associate Professor in the department of Emergency Medicine, Jubilee Mission Medical College and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 03/19/IEC/JMMC&RI
Record Dates: First submitted 2020-07-25; First posted 2020-08-26 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Simulation Training
Keywords: ultrasonography; vascular access; phantom model

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The examiners, examinees and statistician would be blinded to the nature of the model.
  The model would be matched in colour shape and size with the commercially available model. The models would be covered by a plastic surgical drape, with a label on top that said model A or model B.
  The models identity would be known only to the team leader. One the coin toss is complete and model allocated, the allocation would be marked unto a sealed envelope which would be opened only after data entry and analysis.
  Any untoward event needing unmasking of the models like damage to the model, warranting replacement was also carried out by the team leader.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model A first and then B (Other): Model A and B would be randomly allotted to commercial model and IDUP. Intervention limb would involve performing on sequentially on the commercial and IDUP, following which a feed back of the candidates would be recorded about their performance on the same with respect to sonological appearance, tactile feedback, artefacts and ease of performing the procedure. Set time points (time to needle tip visualisation, time to puncture) and no of attempts before successful cannulation would be recorded by an assessor on a pre set proforma.
  Interventions: Other: indigenously developed ultrasound phantom (IDUP)
- Model B first and then A (Other): Model A and B would be randomly allotted to commercial model and IDUP. Intervention limb would involve performing on sequentially on the commercial and IDUP, following which a feed back of the candidates would be recorded about their performance on the same with respect to sonological appearance, tactile feedback, artefacts and ease of performing the procedure. Set time points (time to needle tip visualisation, time to puncture) and no of attempts before successful cannulation would be recorded by an assessor on a pre set proforma.
  Interventions: Other: indigenously developed ultrasound phantom (IDUP)

INTERVENTIONS:
Other: indigenously developed ultrasound phantom (IDUP) — Ultrasound phantom model developed in the department of Emergency Medicine of Jubilee Mission Medical College, to train vascular access.
  Other Names: Jubilee Phantom

SUMMARY:
Point of care ultrasound (POCUS) is used ever more increasingly across the emergency medicine departments in India.

Guided procedures like nerve blocks, vascular access, abscess drainage and foreign body exploration are done more conveniently and efficiently utilising visualisation under ultra sonography.

Several training models are available commercially that aids in training the novice and expert in the field alike. The commercially available models are expensive and inaccessible for most, while the utility of POCUS in Emergency Department (ED) is on the rise. This has lead people to experiment with various models for training which ranges from basic gelatin moulds to ballistic gel. There are only a few studies that compare these with the commercially available products for educational purposes.

The home made models are cheaper and more easily procurable for training making it a relatively favourable choice in financially constrained situations. The investigators have been using a gelatine based training model to train their emergency medicine residents for many years. In this study they intend to assess whether their indigenously developed ultrasound phantom model is comparable to commercially available models for vascular access training.They also sought to assess the better preliminary teaching model for ultrasound guided vascular access: in-plane or out-of-plane approach?

ELIGIBILITY:
Inclusion Criteria:

- All the participants of the ultrasound training module who underwent the vascular access course were considered eligible to participate if they consented for the study

Exclusion Criteria:

- Participants of the ultrasound training module who underwent the vascular access course not giving consent to participate or

Participant ultrasound training module who underwent the vascular access course withdrawing consent for using the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Comparative scoring of the two ultrasound phantom models | 6 hours
  Comparison of the two ultrasound model assessed on a five point Likert scale (1- worst score, 5- best score) in terms of resemblance, tactile feed back, artefacts and ease of use done at the end of the study.

SECONDARY OUTCOMES:
Confidence in performing and teaching ultrasound guided vascular access using in plane approach | 6 hours
  Post workshop confidence level change in performing and teaching needle tracking and vascular access, with in plane approach, assessed on a five point Likert scale (1- least confident score, 5- most confident)
Confidence in performing and teaching ultrasound guided vascular access using out of plane approach | 6 hours
  Post workshop confidence level change in performing and teaching needle tracking and vascular access, with out of plane approach, assessed on a five point Likert scale (1- least confident score, 5- most confident)

OTHER OUTCOMES:
Time taken to visualise needle tip and time taken to puncture vessel and draw fluid in out of plane approach and in plane approach | 6 hours
  Time taken to sonologically visualise the cannulating needles tip and time taken to puncture vessel and aspirate fluid in out of plane approach and in plane approach measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Vimal Krishanan S, MD, Study Director — Manipal Academy of Higher education
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: Yes
Participant data abstracted would be shared as excel sheet. The study protocol also would be shared
Supporting Information: Study Protocol
Time Frame: After publication of the results in a journal, the result would be accessible to all, for a duration no less than one year
Access Criteria: google drive link would be shared